CLINICAL TRIAL: NCT01233921
Title: A Preliminary Study to Evaluate the Effects of Palifermin in Patients at Risk of Chronic Graft-versus-host Disease
Brief Title: Palifermin in Preventing Chronic Graft-Versus-Host Disease in Patients Who Have Undergone Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin, Paul (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Martin, Paul, Member, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2437.00; NCI-2010-01711 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Graft Versus Host Disease; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Graft vs Host Disease; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma | interventions — Fibroblast Growth Factor 7; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (palifermin) (Experimental): Patients receive palifermin IV on days 1-3 in the absence of unacceptable toxicity.
  Interventions: Biological: palifermin; Other: flow cytometry; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (no palifermin) (Active Comparator): Patients do not receive palifermin.
  Interventions: Other: flow cytometry; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: palifermin — Given IV
  Other Names: growth factor, recombinant human keratinocyte; Kepivance; keratinocyte growth factor, recombinant human; recombinant human keratinocyte growth factor; rhKGF
  Arms: Arm I (palifermin)
Other: flow cytometry — Correlative studies
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
RATIONALE: Growth factors, such as palifermin, may prevent chronic graft-versus-host disease caused by donor stem cell transplant.

PURPOSE: This randomized clinical trial studies palifermin in preventing chronic graft-versus-host disease in patients who have undergone donor stem cell transplant for hematologic cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the pharmacodynamic effects of palifermin on thymic function in patients at risk of chronic graft-vs-host disease (GVHD).

II. To evaluate the tolerability of palifermin in patients at risk of chronic GVHD.

OUTLINE: Patients are assigned to 1 of 2 groups based on whether they wish to receive palifermin or not.

GROUP 1: Patients receive palifermin intravenously (IV) on days 1-3 in the absence of unacceptable toxicity.

GROUP 2: Patients do not receive palifermin.

After completion of study treatment, patients are followed up on days 7, 14, 21, and 28.

ELIGIBILITY:
Inclusion Criteria:

* Survival for more than 60 days after an allogeneic hematopoietic cell transplantation (HCT) with growth-factor mobilized blood cells
* Current dose of prednisone at =< 0.5 mg/kg or equivalent or no systemic glucocorticoid treatment
* Ability to remain under care at the Seattle Cancer Care Alliance (SCCA) for at least 28 days after enrollment in the study
* Able and willing to give informed consent

Exclusion Criteria:

* Presence of generalized rash involving more than 50% of the body surface
* Prior diagnosis of chronic GVHD requiring systemic immunosuppressive treatment
* Any prior local irradiation to a field that included the thymus (total body irradiation is allowed)
* History of thymectomy
* Use of rabbit antithymocyte globulin in the pretransplant conditioning regimen
* Use of a graft depleted of T cells
* Any evidence of recurrent or persistent malignancy after HCT
* Participation in another study with chronic GVHD as the primary endpoint
* Any prior history of carcinoma
* Any infection that is not improving during appropriate treatment
* History of palifermin intolerance
* A positive pregnancy test (women of child-bearing potential)
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Martin, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between Nov 2010 and June 2012 during outpatient follow-up after allogeneic hematopoietic cell tranpslantation.
Period: Overall Study
Arm/Group | Arm I (Palifermin) | Arm II (no Palifermin)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Palifermin) | Arm II (no Palifermin) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13) | 41 (11) | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Number of Recent Thymic Emigrants (RTE) Cluster of Differentiation (CD)4 T Cells in the Blood
Description: RTE CD4 T cells will be defined according to co-expression of CD3, CD4, CD31, CD45RA, and CCR7. Cells will be counted by flow cytometry at baseline and at 4 weeks and changes will be measured as cells per microliter of blood. Positive results indicate an increase in the number of cells between baseline and 4 weeks. Negative results indicate a decrease in the number of cells between baseline and 4 weeks.
Time Frame: Baseline and 4 weeks after administration of palifermin
Measure: Mean (Standard Deviation); unit: cells per microliter of blood
Arm/Group | Arm I (Palifermin) | Arm II (no Palifermin)
Number analyzed (Participants) | 3 | 3
cells per microliter of blood | -2 (3) | -22 (51)

2. Secondary Outcome: Changes in the Number of Naive CD4 T Cells in the Blood
Description: Naive CD4 T cells will be defined according to co-expression of CD3, CD4, CD45RA, and CCR7. Positive results indicate an increase in the number of cells between baseline and 4 weeks. Negative results indicate a decrease in the number of cells between baseline and 4 weeks.
Time Frame: Baseline and 4 weeks after administration of palifermin
Measure: Mean (Standard Deviation); unit: cells per microliter of blood
Arm/Group | Arm I (Palifermin) | Arm II (no Palifermin)
Number analyzed (Participants) | 3 | 3
cells per microliter of blood | -3 (4) | -25 (58)

ADVERSE EVENTS:
Arm/Group | Arm I (Palifermin) | Arm II (no Palifermin)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Palifermin) (N=3) | Arm II (no Palifermin) (N=3)
rash (Skin and subcutaneous tissue disorders) | 2 | 1
pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
oral mucosal change (Gastrointestinal disorders) | 3 | 0 — Hyperkeratosis and taste changes
pain (Musculoskeletal and connective tissue disorders) | 2 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
edema (General disorders) | 1 | 0
anorexia (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 2 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes